CLINICAL TRIAL: NCT05768061
Title: HBV Reactivation in Anti CD20 Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Rawi Hazzan, Head of liver unit, HaEmek Medical Center, Israel
Other Study IDs: 0122-21-COM2
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hepatitis B
Keywords: anti CD20; Rituximab; HBV- hepatitis B virus
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to test and describe the frequency of hepatitis B virus reactivation in patients who received anti-CD20 drugs for a wide variety of autoimmune and hemato-oncological diseases in order to find out whether a group of patients from a certain field was more sensitive to treatment in this respect than patients from other fields.

DETAILED DESCRIPTION:
Hepatitis B virus(HBV) is the most common chronic virus worldwide. it causes an infection of the liver (hepatitis B) and it is transmitted from person to person through contact with virus-contaminated blood, through sexual intercourse, and vertically from mother to fetus.

Anti CD20 drug or Rituximab is an anti-CD20 monoclonal antibody on the surface of B lymphocytes, which induces cell death (apoptosis) and thus causes depletion. The main side effects of rituximab are infectious and hypersensitivity reactions. It can also increase the chance of hepatitis B reactivation to the point of acute hepatitis.

The information for this retrospective study will be collected from clalit health care's databases.

The patients will be sorted according to the indications for which the treatment with anti-CD20 drugs was given in order to see the differences in the response to the drug in different groups of patient

ELIGIBILITY:
Inclusion Criteria:

* subjects (men and women) of age 18 and above, who received anti-CD20 (Rituximab) drugs as a treatment for a variety of diseases .

Exclusion Criteria:

* healthy subjects.
* subjects under the age 18.
* subjects who did not receive anti CD20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of subjects who received anti-CD20 drugs as a treatment for a variety of diseases between the years 2000 to 2021, within Clalit Health care record database.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
HBV DNA in the blood. | about 10 minutes per blood test.
  Reactivation of HBV is defined when one of these three conditions exist:
  1. when Participant has An increase of more than log1 in the concentration of HBV DNA in the blood.
  2. when Participant has A positive HBV DNA result compared to a negative result before starting treatment with Rituximab (anti CD20).
  3. when Participant has HDV (hepatitis D virus) DNA result greater than 20000 IU/mL in the absence of a test before starting treatment
     * The HBV DNA concentration at the beginning of the treatment was defined in the time period between six months before the start of the treatment and 30 days after the start of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rawi Hazzan, MD, Principal Investigator — haemek medical center
Locations (1):
- HaEmek Medical Center, Afula, Northern District, Israel